CLINICAL TRIAL: NCT05984004
Title: A Double-blind, Randomized, Placebo-controlled Study to Evaluate the Safety of Postbiotic Nasal Spray Using Killed Spores of Bacillus Subtilis DSM32444 in Healthy Volunteers
Brief Title: Safety Evaluation of Intranasal Use of DSM 32444 Postbiotic in Humans
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Huro Biotech Joint Stock Company (Industry)
Collaborators: Thai Binh University of Medicine and Pharmacy (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HSP32444.01
Record Dates: First submitted 2023-07-31; First posted 2023-08-09 (Actual); Last update posted 2024-04-12 (Actual); Status verified 2024-04

CONDITIONS: Rhino Sinusitis
Keywords: Acute Rhinosinusitis; Chronic Rhinosinusitis; Allergic Rhinosinusitis
MeSH Terms: conditions — Rhinosinusitis; Rhinitis, Allergic, Perennial | interventions — Saline Solution

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (Placebo Comparator): Healthy volunteers in Control group receives a nasal spray containing 0.9% NaCl isotonic saline solution.
  Interventions: Drug: 0.9% NaCl isotonic saline solution
- SPEROVID (Experimental): Healthy volunteers in SPEROVID group receives a nasal spray containing inactivated Bacillus subtilis DSM32444 (postbiotic)
  Interventions: Combination Product: Bacillus subtilis DSM32444, inactivated

INTERVENTIONS:
Drug: 0.9% NaCl isotonic saline solution — The placebo-control in the phase I study was a 0.9% NaCl isotonic saline solution. This nasal spray solution has no pharmacological effect, but is considered to have a cleansing effect on the nose, supporting the treatment of nasal symptoms in nasal pathology. The solution is prepared by extracting 5 mL from 0.9% NaCl intravenous infusion 500 mL PP bottle (B.Braun, Germany, product declaration No. VD-32732-19). The solution is bottled in the same fully-sealed nasal spray device containing Bacillus subtilis DSM 32444 postbiotic, used for Sperovid.
  Other Names: 0.9% NaCl
  Arms: Control
Combination Product: Bacillus subtilis DSM32444, inactivated — Postbiotic DSM32444 is manufactured by HURO BIOTECH Company as a drug-grade active pharmaceutical ingredient. The Class A medical device containing Postbiotic DSM32444 is called Sperovid, which is manufactured by Dong Duoc Viet under ISO 13485:2016 standards for medical device. Sperovid has registration number: 220000033/PCBA-LA
  Other Names: Sperovid, Speromed, Sperokid, SPOR-COV
  Arms: SPEROVID

SUMMARY:
Rhinitis is a type of upper respiratory infection with a common nasal pathology especially in Southeast Asia, which is characterized by the presence of one or more of the following symptoms: itchy nose, sneezing, runny nose, and nasal congestion. The treatment of acute rhinosinusitis and allergic rhinitis in hospitals is currently carried out according to the general professional guidance of the Vietnam Ministry of Health. A common treatment regime for patients with rhinosinusitis in Vietnam includes a combination of steroids and antibiotics (Neomycin/Dexamethasone/ Xylometazoline) administered as a nasal spray, in adjunct with Amoxicillin/clavulanate 875/125 mg taken orally every 12- hours. The duration of treatment for patients is about 10 days depending on the severity of the disease. During the treatment period, a change in the systemic antibiotic regimen is necessary if the observations after 3 to 5 days of treatment do not show signs of a satisfactory response.

Current concerns about antimicrobial resistance (AMR) as well as side effects of corticosteroids and antihistamines have led to an urgent need for a naturebased next generation therapeutic approach that is safe, effective and helps in addressing the issues of AMR.

There have been multiple research studies supporting the efficacy of bacterialbased approaches in the prevention of viral respiratory infections, and that have potential for treatment. For use in the respiratory tract, it is necessary to have a completely sterile product to ensure safety in the long-term and there is a need for safety assessment of products both in animal models and human studies.

This phase of the study aims to evaluate the safety in humans of a nasal spray using a postbiotic preparation of Bacillus subtilis DSM32444 and that is a sterile inert bioparticle.

DETAILED DESCRIPTION:
Rhinitis is a type of upper respiratory infection and a common nasal pathology especially in Southeast Asia, which is characterized by the presence of one or more of the following symptoms: itchy nose, sneezing, runny nose, and nasal congestion. Other symptoms occasionally experienced include headache, excessive pain reaction, cough, fever. Rhinitis can be idiopathic or due to a variety of causes, including allergens, medications, endocrine/metabolic, infectious, inflammatory, and abnormal nasal structures. Rhinosinusitis in general is not a dangerous pathological condition, however the frequency of the disease is relatively high with statistics showing that all people experience it at least once in their lives. Common rhinosinusitis symptoms include severe facial pains and difficulties in breathing. Hence, most patients are prescribed corticosteroids, antihistamines, and antibiotics for immediate decongestion and anti-inflammatory effects. Current concerns about antimicrobial resistance (AMR) as well as the documented side effects of corticosteroid and antihistamine have led to an urgent need for a nature-based next generation therapeutic approach that is safe, effective and helps in addressing AMR problem. Preclinical studies of inactivated Bacillus subtilis strain DSM32444 conducted by collaborating UK universities and laboratories have shown potential therapeutic benefits with anti-inflammatory mechanisms that may be useful in other viral infections of the respiratory tract. The reason for using an inactivated spore is because various publications have identified risks of inhalation of high doses of live bacteria in the respiratory tract and lungs. DSM32444 also carries GRAS status for human use. An accredited, cGLP, repeat-dose toxicology study also confirmed complete safety in rodent models after high doses of treatment.

The investigators think there is a likelihood to apply this postbiotic technology to mitigate the overuse of antibiotics, corticosteroids, and antihistamines. The aim of this study is to evaluate the safety nasal spray using the postbiotic Bacillus subtilis DSM32444 when used in humans.

* Study population: Sample size for Phase 1 is 60 healthy volunteers to assess tolerance.
* Description of Sites: the study is carried out at Thai Binh University of Medicine and Pharmacy and Thai Binh University of Medicine and Pharmacy Hospital.
* Description of Study intervention:

The Phase I study is a double-blind, parallel-group, randomized, placebo controlled study. Study participants who are healthy volunteers were randomly assigned 1:1 to either the postbiotic DSM32444 nasal spray (SPEROVID) or the placebo (0.9% NaCl). Study subjects who are healthy volunteers, confirmed by routine physical examination of the research facility, will be invited to participate in the phase I study. The randomization is carried out according to the 4-block strategy using envelopes with predetermined random codes. Study subjects will be given codes in turn sealed in sequentially numbered envelopes. The research product is prepared in a double-blind form, on the label there are random codes matching the code assigned to the study object. The duration of the study regimen is 7-days, except for early withdrawal from the study for safety reasons. The research product (SPEROVID or placebo) is nasally administered as a spray 2-3 times daily, with each administration being 0.1ml/nostril (total 0.2 mL/administration). Researchers will follow up with volunteers for safety evaluation of the products, analysis of the subject's complaints of disease and other special issues (if applicable), physical examination and laboratory tests. If any adverse events are detected, the investigator should immediately record the information in the source literature and CRF, specifying the nature of the AE, the duration of the AE, and other characteristics.

* The study data after collection will be analyzed statistically using SAS 9.4. The normal distribution of statistical samples will be evaluated by the Kolmogorov- Smirnov-Lilliefors test, the uniformity of variance will be verified by Levene's test. The continuous variables will be analyzed using a two-dimensional variance test or covariance analysis (ANOVA/ANCOVA) in the case of a normal distribution and using the ANOVA non-parametric Kruskal-Wallis test in the case of a non-standard distribution. Repeatable measurement analyses will be used where appropriate. Differences between treatment groups in terms of duration of major symptoms of acute respiratory infection and average time to resolution will be assessed using the Student's t-test or the Mann-Whitney test. Chi-Square (or Fisher's exact test) will be used to evaluate the difference between the ratios. Analysis of classification data is carried out using the Cochran-Mantel Haenszel test. In the absence of further note, the continuous variables are expressed by the mean ± standard deviation. The Cox analysis model and log-rank testing will be used to compare variables of the time type leading up to an event.
* Expected outcomes: The nasal spray using postbiotic Bacillus subtilis DSM32444 (SPEROVID) is safe and well tolerated among healthy volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers must be ≥18 years of age, at the time of signing the informed consent.
* Participants who are able to use an e-Diary or Paper Diary during the study to report their health status
* Participants capable of giving a signed informed consent form (ICF)

Exclusion Criteria:

* Planned travel outside of the study area during the study period.
* Use of any investigational drug within 30 days prior to Day screening. No investigational products are permitted for use during the conduct of this study
* A known history of alcohol or drug abuse within the last 2 years
* Existence of any medical condition, which in the opinion of the investigator, might significantly affect the subject's ability to complete this trial; or their safety in this trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2022-09-26 (Actual); Primary Completion 2022-11-22 (Actual); Study Completion 2023-04-20 (Actual)

PRIMARY OUTCOMES:
To compare the safety and tolerability following multiple doses of postbiotic DSM32444 nasal spray for 7 days with Placebo in Heathy Volunteers | Day 1 to Day 7
  * Incidence of Adverse Events (Nasal Congestion, Itchy Nose, Allergic Reaction/Rash, Sneezing, Nasal Discharge, Weeping, Itchy eyes, Itchy ears, Sore throat, Nausea/Vomiting)
  * Incidence of Serious Adverse Events (Adverse events leading to discontinuation of study products, Adverse events leading to withdrawal of subjects from the study, Deaths up to the time of study data cut off)
  * Incidence of Related Adverse Events
  * Incidence of Related Serious Adverse Events

CONTACTS AND LOCATIONS:
Overall Officials: Kien T NGUYEN, PhD, Principal Investigator — Thai Binh University of Medicine and Pharmacy
Locations (1):
- Thai Binh University of Medicine and Pharmacy, Thái Bình, Thai Binh, Vietnam

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Baraniuk JN. Pathogenic mechanisms of idiopathic nonallergic rhinitis. World Allergy Organ J. 2009 Jun 15;2(6):106-14. doi: 10.1097/WOX.0b013e3181aadb16. PMID 24229057
- [Background] James J, Meyer SM, Hong HA, Dang C, Linh HTY, Ferreira W, Katsande PM, Vo L, Hynes D, Love W, Banyard AC, Cutting SM. Intranasal Treatment of Ferrets with Inert Bacterial Spores Reduces Disease Caused by a Challenging H7N9 Avian Influenza Virus. Vaccines (Basel). 2022 Sep 19;10(9):1559. doi: 10.3390/vaccines10091559. PMID 36146637
- [Background] Wallace DV, Dykewicz MS, Bernstein DI, Blessing-Moore J, Cox L, Khan DA, Lang DM, Nicklas RA, Oppenheimer J, Portnoy JM, Randolph CC, Schuller D, Spector SL, Tilles SA; Joint Task Force on Practice; American Academy of Allergy; Asthma & Immunology; American College of Allergy; Asthma and Immunology; Joint Council of Allergy, Asthma and Immunology. The diagnosis and management of rhinitis: an updated practice parameter. J Allergy Clin Immunol. 2008 Aug;122(2 Suppl):S1-84. doi: 10.1016/j.jaci.2008.06.003. No abstract available. PMID 18662584
- [Background] Huang JM, La Ragione RM, Nunez A, Cutting SM. Immunostimulatory activity of Bacillus spores. FEMS Immunol Med Microbiol. 2008 Jul;53(2):195-203. doi: 10.1111/j.1574-695X.2008.00415.x. Epub 2008 Apr 21. PMID 18430003